CLINICAL TRIAL: NCT03979534
Title: Protecting Kidneys Through a Low Protein Diet: A Stepwise Multiple-Choice System Approach
Acronym: ProReRePro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHM-2016-S8/05
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Diseases
Keywords: low-protein diet; pre-dialysis; chronic kidney disease; nutritional care; start of dialysis; incremental dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet group (Experimental): Diet follow-up to personalize a low-protein diet for each patient. All patients following a low protein diet one month or more compose the "diet group".
  Interventions: Other: low protein diet
- Control group (No Intervention): Patients who accepted to take part of the study but refused the low protein diet and patients who discontinued the diet on the first month compose the control group.

INTERVENTIONS:
Other: low protein diet — Patients will be managed with a restricted protein intake (controlled protein diets with a mean target at 0.6 g / kg / day of protein, according to a choice of dietary approaches, adapted to the situation of each patient).
  Arms: Diet group

SUMMARY:
Nephrology care continues to progress and recommendations are now focused on delaying as much as possible the need for renal replacement therapy ("intent-to-defer"strategy). Protein restriction is a valuable tool for stabilizing chronic kidney disease (CKD) and retarding the need for renal replacement therapy, but the best diet to be prescribed is still matter of discussion. This study is aimed at identifying implementation strategies for nutritional management of advanced CKD.

DETAILED DESCRIPTION:
The recent paradigm on dialysis start suggests that an intention to defer policy should be preferred to beginning dialysis early ("the earliest the best" strategy). This strategy is further supported by the consideration that patient profiles are changing with the increasing proportion of older and higher comorbidity patients. In high comorbidity patients, survival is not necessarily improved by dialysis.

Nutritional care, adapted to each patient's needs and preferences, could in part answer these demands. Indeed, renal function has a strict correlation with dietary patterns. Low protein diets may have two favourable effects: 1) slowing down kidney function decline and 2) delaying the need of replacement therapy (metabolic stabilizing). In dialysis, the nutritional state is the most important survival indicator, and nutritional follow-up should allow starting dialysis in a good nutritional status.

The study proposed here is an implementation study with a principal aim to improve the use of low protein diets in the clinical setting, by offering a multiple choice approach and by adapting the diets to the patients' needs.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients followed on the unit for advanced CKD, with Kidney disease stage 4-5 or stage 3 with fast progression and without contraindications.

Exclusion Criteria:

* Malnutrition or short life-expectancy
* Patients aged less than 18 years old
* Pregnant women,
* Incapacity to complete the free-consent form,
* Pateints refusing participation in the study,
* Patients without healthcare coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-04-02 (Estimated); Study Completion 2023-04-02 (Estimated)

PRIMARY OUTCOMES:
Adherence to the multiple-choice diet program | 4 years
  Percentage of patients who drop-out of the multiple choice diet program

SECONDARY OUTCOMES:
Kidney survival | 4 years
  The "kidney survival" from the beginning of the diet to the start of renal replacement therapy
Patient survival | 4 years
  The patient survival compared to reference data (from the Réseau Epidemiologie, Information, Néphrologie) and international registers.
Cost of the treatment | 4 years
  Cost of the treatment, including diet, renal replacement therapy and pharmacological interventions.
Patients included in a transplantation program | 4 years
  Percentage of patients without contraindications enrolled on the pre-emptive kidney transplant list.
Patients included in a home dialysis program | 4 years
  Percentage of patients without contraindications who started a home dialysis treatment
Patients included in an incremental dialysis program. | 4 years
  Percentage of patients without contraindications who started dialysis with an incremental schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgina Piccoli, MD, Principal Investigator — Centre Hospitalier le Mans
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No